CLINICAL TRIAL: NCT02545426
Title: Myocardial Stunning During Hemodialysis: Role of Dialyste Calcium Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rosilene Motta Elias Coelho, M.D., Ph.D., University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Myocardial stunning - Calcium
Record Dates: First submitted 2014-08-17; First posted 2015-09-10 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Myocardial Stunning; End-stage Renal Disease
Keywords: myocardial stunning; dialysate calcium concentration; nutritional status; hemodinamic; hemodialysis
MeSH Terms: conditions — Myocardial Stunning; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium dialysate 2.5mEq/L (Active Comparator): Dialysis with low calcium concentration
  Interventions: Other: Change the dialysate calcium concentration
- Calcium dialysate 3.5mEq/L (Active Comparator): Dialysis with high calcium concentration
  Interventions: Other: Change the dialysate calcium concentration

INTERVENTIONS:
Other: Change the dialysate calcium concentration — The dialysate calcium concentration will be changed according to the prior concentration

SUMMARY:
Chronic kidney disease (CKD) is linked to elevated mortality rate, and cardiovascular disease is the main cause related to this outcome. The cardiovascular mortality among patients on conventional hemodialysis (CHD) is high, achieving up to 30 times more risk of death when comparing to individuals of same age on general population. Congestive heart failure can develop in 25% to 50% of patients, leading to a worse prognosis. CKD patients present anatomic and functional abnormalities on peripheral bed vases and also cardiovascular abnormalities that can cause myocardial ischemia. This last usually is transitory and lead to left ventricular dysfunction that can persist even after the end of dialysis session despite normal coronary perfusion. The prolonged dysfunction is called myocardial stunning (MS). Patients on CHD are subject to hemodynamic instability, myocardial ischemia and development of regional abnormalities of myocardial wall (ARPM´s). MS induced by intradialytic ischemia is a complication that can be minimized by applying techniques associated to more stability during the CHD, as cool dialysate or increasing the length of the therapy. The goal of the present study is to evaluate the behavior of cardiovascular system (trough hemodynamic performance during CHD, accessing MS by echocardiography technique, and biomarkers associated to MS). Finally, the investigators aimed to investigate the role of two different dialysate calcium concentration (2,5 and 3,5 mEq/l) in the genesis of MS during CHD. The elucidation of pathogenesis of MS during CHD might help us modified hemodialysis technique in order to prevent MS, and reduce the high cardiovascular mortality among CKD patients.

DETAILED DESCRIPTION:
Patients on hemodialysis patients present anatomic and functional abnormalities on peripheral bed vases and also cardiovascular abnormalities that can cause myocardial ischemia. This last usually is transitory and lead to left ventricular dysfunction that can persist even after the end of dialysis session despite normal coronary perfusion. The prolonged dysfunction is called myocardial stunning (MS). Patients on dialysis are subject to hemodynamic instability, myocardial ischemia and development of regional abnormalities of myocardial wall (ARPM´s). Some authors have demonstrated that CHD cause segmental and global myocardial ischemia, and up to 65% of patients have recurrent myocardial ischemia. There are some associated factors: high ultrafiltration rates, intradialytic hypotension, reduced systolic blood pressure and high risk of cardiovascular events and death. MS induced by intradialytic ischemia is a complication that can be minimized by applying techniques associated to more stability during the CHD, as cool dialysate or increasing the length of the therapy. More specifically, MS can be the result of repair process, with oxygen free radicals generation and reduction of the synthesis of contractile proteins, in association with a reduced muscle responses to calcium which in turns lead to ventricular dysfunction (the calcium hypothesis). The goal of the present study is to evaluate the behavior of cardiovascular system (trough hemodynamic performance during CHD, accessing MS by echocardiography technique, and biomarkers associated to MS). Finally, the investigators aimed to investigate the role of two different dialysate calcium concentration (2,5 and 3,5 mEq/l) in the genesis of MS during CHD. The elucidation of pathogenesis of MS during CHD might help us modified hemodialysis technique in order to prevent MS, and reduce the high cardiovascular mortality among CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on conventional hemodialysis

Exclusion Criteria:

* Congestive heart failure, arrhythmia, active infection, cancer

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
myocardial stunning diagnosis by echocardiography technique strain | 1 week
  Investigate the role of two different dialysate calcium concentration (2,5 and 3,5 mEq/l) in the genesis of myocardial stunning diagnosis by echocardiography technique strain

CONTACTS AND LOCATIONS:
Overall Officials: Rosilene M Elias, M.D., Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil